CLINICAL TRIAL: NCT01929954
Title: Phase 1/2, Randomized, Controlled Assessment of the Safety Of Gintuit™ Versus Bio-Gide® in Subjects Requiring Socket Grafting
Brief Title: Safety Study of Gintuit™ in Subjects Requiring Socket Grafting
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Changes in corporate business environment
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-PER-005-GT
Record Dates: First submitted 2013-08-13; First posted 2013-08-28 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gintuit (Experimental): Subjects with a posterior tooth (molar or premolar) socket created by atraumatic extraction will be grafted with freeze-dried bone allograft (ie, MinerOss™). The primary wound bed will consist of exposed alveolar bone and bone graft imbedded in coagulum of blood from the socket for both treatments. The test treatment GINTUIT will be inlayed within the defect over the socket graft material, and stabilized with resorbable tacking sutures. An additional single layer of GINTUIT will cover the entire surface of the extraction socket at approx. 2-3 mm beyond the margins of the wound and fixed with non-resorbable sutures. The lower layer of this additional layer should be in contact with the previously applied GINTUIT.
  Interventions: Biological: Gintuit
- Bio-Gide (Active Comparator): Subjects with a posterior tooth (molar or premolar) socket created by atraumatic extraction will be grafted with freeze-dried bone allograft (ie, MinerOss™). The primary wound bed will consist of exposed alveolar bone and bone graft imbedded in coagulum of blood from the socket for both treatments. The control treatment will be a collagen membrane (ie, Bio-Gide, applied per the Package Insert) inlayed within the defect over the socket graft material, and stabilized with resorbable tacking sutures. Crossed suspensory type sutures should also be placed over Bio-Gide, depending on the degree of stabilization needed. In all subjects, care should be taken in suturing to avoid advancement of the buccal gingival flap.
  Interventions: Device: Bio-Gide

INTERVENTIONS:
Biological: Gintuit — One time placement of Gintuit over socket graft.
  Arms: Gintuit
Device: Bio-Gide — One time placement of Bio-Gide over socket graft.
  Arms: Bio-Gide

SUMMARY:
This is a prospective, randomized, controlled, parallel group Phase 1/2 assessment of the safety of GINTUIT versus Bio-Gide in subjects who have a posterior tooth requiring extraction. The incidence and severity of adverse events will be summarized by group (GINTUIT and Bio-Gide).

DETAILED DESCRIPTION:
This study will evaluate the safety of GINTUIT as compared with Bio-Gide in subjects who have a posterior tooth requiring extraction. The use of GINTUIT in this investigational clinical indication may eliminate/reduce the need for aggressive flap advancement with its concomitant morbidity, while, at the same time, obtaining stable closure over a grafted socket. It is anticipated that GINTUIT will facilitate tissue granulation, followed by tissue coverage with site appropriate tissue (ie, keratinized tissue) that is needed for long term stability of the final restoration.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age but no more than 75 years of age.
* Subject has a posterior (molar or premolar) socket created by atraumatic extraction with a post extraction socket of a minimum of 5 mm in both the mesial-distal (M-D) and buccal-lingual (B-L) dimensions that requires bone grafting.
* Subject has sufficient buccal bone plate at the site of the planned tooth extraction (ie, the residual socket should be of a form that would retain bone graft material), as judged by the Principal Investigator.
* Females of childbearing potential must have a documented negative urine pregnancy test. All subjects must agree to use acceptable methods of contraception for the duration of the study.
* Subjects must have read, understood, and signed an institutional review board (IRB)-approved Informed Consent Form (ICF).
* Subjects must be able and willing to comply with protocol requirements.

Exclusion Criteria:

* Subject with any systemic conditions that could compromise wound healing and preclude periodontal surgery (ie, bleeding disorder, cancer, except localized basal cell or squamous cell cancer of the skin with no metastasis; human immunodeficiency virus; or bone metabolic diseases [ie, osteoporosis or Paget's disease]).
* Subject who is currently receiving, anticipates receiving or has received within 30 days prior to Day 0: inhaled or systemic corticosteroids (ie, oral, IV), immunosuppressive agents or radiation therapy, and/or chemotherapy, which could compromise wound healing and preclude periodontal surgery.
* Subject who has had oral/periodontal surgery within 30 days prior to Day 0 or anticipates having oral/periodontal surgery within 30 days after Day 0.
* Subject with acute mucosal infection, including suppuration or induration in the area of intended surgery.
* Subject, who in the opinion of the Principal Investigator, will require a sinus lift procedure to place dental implants in the surgical area.
* Subject without at least 1 tooth adjacent to the area to be treated.
* Subject has a history of alcohol or substance abuse within the previous 12 months of Screening that could interfere with study compliance or protocol requirements.
* Subject who has used any tobacco product within 6 months of Screening.
* Subject with known hypersensitivity to porcine or bovine collagen, gentamicin or surfactants.
* Subject who has received an investigational drug, device, or biological/bioactive treatment within 30 days prior to Day 0 (medical or dental).
* Subject who was previously treated with Gintuit, or any other cell therapy at the target treatment site or immediately adjacent teeth.
* Female subject that is lactating.
* Subject, who in the opinion of the Principal Investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 12 months post treatment

SECONDARY OUTCOMES:
Optimal product configuration (ie, single, folded, or z-folded) | One month after placement of Gintuit in the last subject in the last successful cohort
  Subjective assessment based on the results of the analyses of safety, efficacy and product handling (from surgeon input) data
Number of participants reporting loose graft material | Up to 21 days post treatment
Percentage of participants with soft tissue closure | Up to 4 weeks post treatment
Measurements of bone height | Up to 6 months post treatment
Gintuit product handling | At Day 0
  Rated as excellent, very good, good, adequate, poor
Number of participants with visible loss of graft material | Up to 3 months post treatment
Percentage of participants with convex, normal and concave soft tissue contour | Up to 6 months post treatment
Measurement of soft tissue ridge contour | Up to 6 months post treatment
Measurement of soft tissue thickness | Up to 6 months post treatment
Percentage of participants with color and texture match | Up to 6 months post treatment
Percentage of participants with a clinically significant physical reduction of crestal ridge height | Up to 6 months post treatment
  Clinically significant defined as > 2 mm loss at the crest of the ridge at the graft site compared to Day 0
Measurements of soft tissue ridge height | Up to 6 months post treatment
Measurements of ridge width of hard tissue | Up to 6 months post treatment
Bone quality | Up to 6 months post treatment
  Regularity and density of the cortical and trabecular bone using the system described by Norton and Gamble (Quality Levels 1, 2/3, 4 and 4 (failure zone))
Percentage of participants with acceptable implant stability | Up to 12 months post treatment
  Acceptable implant stability defined as an implant stability quotient of >/= 55

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G. Murphy, DDS, MS, Principal Investigator — Kevin G. Murphy Associates, P.A.
Locations (1):
- Kevin G. Murphy and Associates, P.A., Baltimore, Maryland, United States